CLINICAL TRIAL: NCT03213392
Title: Enzymatic Evaluation of General Anesthetic Induced Neurotoxicity in Patients With Aneurysmal Subarachnoid Haemorrhage
Brief Title: Enzymatic Evaluation of General Anesthetic Induced Neurotoxicity in Patients With Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Mukilan Balu (Other)
Responsible Party: Sponsor-Investigator, Mukilan Balu, principal investigator-resident in the department of neuroanesthesia, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Other Study IDs: NK/2677/DM/351
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Anesthetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — serum from blood samples and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SUPRA ORBITAL KEYHOLE CLIPPING/ COILING: Aneurysms should be either clipped or coiled to prevent re rupture general anesthesia is required to carry out these procedures.various anesthetic agents are used as an maintenance agents.
  Interventions: Drug: Anesthetic Agents

INTERVENTIONS:
Drug: Anesthetic Agents — four different anesthetic agents will be used during the surgical clipping or coiling of the aneurysm for the maintenance of anesthesia.
  Other Names: ANESTHETIC AGENTS FOR MAINTENANCE OF SURGERY

SUMMARY:
General anesthetic induced neurotoxicity has received considerable attention in the past decade from various pre-clinical studies in rodents and non-human primates. Which demonstrated that exposure to general anesthetic agents for a longer duration can induce neuronal cell death that can lead to adverse neurodevelopmental outcomes.

The neuroapoptosis and impairment of neurodevelopmental processes has been postulated as the underlying mechanism, but the molecular mechanisms was not completely understood. Various hypothesis has been proposed they are- Antagonistic effect on N-methyl-D-aspartate receptors and agonistic effect on gamma-aminobutyric acid type A receptors; mitochondrial perturbations and activation of reactive oxygen species and dysregulation of intracellular calcium homeostasis. They trigger neuroapoptosis and cell death through the activation of caspases.3 Caspases, a group of cysteine proteases, plays an important role in regulation and execution of apoptosis. Caspase-3 is most important since it is activated by many cell death signals and cleaves a variety of important cellular proteins.4 Various anesthetic agents like isoflurane, halothane, sevoflurane, nitrous oxide and propofol causes neurotoxicity by activation of caspase-3. Which has been proven from various animal studies western blot analysis, immunohistochemical analysis and flow cytometric analysis.3, 5-9 Though it is documented that exposure to general anesthetics causes neurotoxicity during active brain growth in animals, there is no evidence of such effects in adult humans.10 and it is difficult to separate the effects of anesthetics from surgical impact and other factors associated with diseases.11 The patients with aneurysmal subarachnoid hemorrhage (SAH) have variable degree of neurological insults and it is possible, based on the evidence from animal models that administration of general anesthetics could add to the neuronal insults.

DETAILED DESCRIPTION:
Sixteen patients will be included for the study under each intervention (surgery or endovascular coiling). Total thirty two patients who meet the inclusion criteria will be recruited to the study. The patients will be randomized into four groups to receive Propofol (Group P), Isoflurane (Group I), Sevoflurane (Group S) or Desflurane (Group D) using a computer generated algorithm for the maintenance of anesthesia.

The surgery or endovascular coiling will be conducted by an experienced neurosurgeon or radiologist who will be blinded to the anesthetic agent used for maintenance of anesthesia. Pre-anesthetic checkup will be conducted prior to the intervention. Patient will be thoroughly examined and all the investigations will be reviewed. Written informed consent will be obtained from the patient's next of kin.

ANESTHESIA PROTOCOL:

Routine non-invasive monitors will be attached to the patients. It will include noninvasive blood pressure (NIBP), heart rate (HR), electrocardiography (ECG), pulse oximetry (SpO2), end tidal carbon dioxide (EtCO2), state entropy (SE) and urine output. All patients will be preloaded with 10-15 ml/kg of normal saline Fentanyl will be administered intravenously in dose of 2µg/kg prior to induction followed by 0.5-2 µg/kg/hr as infusion. Patients in all 4 groups will be induced with propofol 1 to 2 mg/kg, titrated to loss of verbal response. Vecuronium 0.1 mg/kg will be given to facilitate tracheal intubation. Lignocaine 1.5mg/kg will be given 120 seconds prior to laryngoscopy. For beat to beat monitoring of blood pressure and blood gas analysis an arterial catheter will be placed after induction of anesthesia. Patients will be maintained according to the group allocation along with 50/50% Oxygen/Air. BIS monitoring will be used to maintain comparable depth of anesthesia in all the groups and will be titrated to keep SE in range of 40 to 60. Vecuronium will be given intermittently to maintain less than two twitches on neurostimulation. Body temperature will be maintained using forced air warming blanket.

Normal Saline will be used as the intraoperative fluid. PaCO2 will be maintained around 32-36 mmHg. Neuromuscular blockade will be reversed with a combination of neostigmine 50 µg /kg and glycopyrrolate 10 µg /kg. Subsequently trachea will be extubated.

The patients who cannot be extubated will be shifted to neurosurgical intensive care unit for elective ventilator support.

Intra-operatively hemodynamic monitoring, temporary clipping time and any incidence of aneurysm rupture will be noted. Brain bulge at the time of dural reflection will be noted. Patient status will be assessed at the end of surgery in terms of extubation and neurological status i.e. GCS.

STUDY VARIABLES -

PREOPERATIVE:

Demographic data of the patient, day of ictus, day of admission in hospital, day of surgery, WFNS, Fischer grades and any comorbidities will be noted. Neurological examination including the GCS and presence or absence of any preoperative neurological deficit will also be noted.

INTRA OPERATIVE:

Heart rate (HR), systolic blood pressure (SBP), mean arterial pressure (MAP), pulse oximetry (SpO2) , temperature and end tidal carbon dioxide (EtCO2) will be noted at the time of induction, intubation, incision, application of head pins, bone flap reflection, Dural reflection, clipping, Dural closure, skin closure and prior to cessation of anaesthesia. Patients heart rate and blood pressure will be kept as close to baseline as possible. Any sustained increase in BP more than 30% of the baseline values will be considered as intra-operative hypertension. Hypotension will be considered if MAP < 70 mmHg or SBP < 90 mmHg. The management of hypertension or hypotension will be at the discretion of the attending anesthesiologist.

The brain relaxation scoring will be done following bone flap reflection using four point scale. The temporary clipping time, intra operative rupture of aneurysm, intra operative intravenous fluid administration, blood loss, urine output will be noted.

PROTOCOL FOR ENZYME STUDY AND ESTIMATION:

Patient's baseline cerebrospinal fluid (CSF) and serum blood sample will be collected. The baseline CSF will be collected via an indwelling lumbar subarachnoid catheter placed prior to intervention as a modality to prevent the complication associated with SAH like vasospasm and to facilitate the drainage of SAH. A venipuncture will be done and 2 to 3 ml of blood sample will be collected in plain vial for serum/EDTA for plasma.The second CSF and serum blood sample will be collected after 1 hours of exposure to anaesthesia. The third sample will be collected following completion of intervention or after the cessation anesthetic agent, whichever is earlier.

Caspase 3 enzyme level would be estimated using a quantitative ELISA kit with precoated antigen wells and known standards by a double antibody sandwich technique.

Sample collection and storage- Blood samples would be collected in plain vials/vacutainers. CSF samples would be collected in cryovials. Blood samples would be allowed to clot at room temperature for 1 hour. The clotted blood in the plain vacutainers would be centrifuged at 2000 rpm for 15 minutes to separate out the serum. Serum would be pipetted off into cryovials. All samples would be stored at -80˚C immediately till further analysis.

Caspase 3 enzyme estimation The following steps will be followed for enzymatic evaluation-

1. The ELISA kit stored at 40C will be taken out of refrigerator 20 minutes before performing the test to equilibrated it to the room temperature.
2. Different concentration of Human-caspase 3 standards with known values and test samples with unknown values would be added to the coated wells in the pre-coated microplate.
3. Biotinylated Human caspase 3 antibody liquid,enzyme conjugate liquid and colour reagent are prepared 30 minutes before use
4. Elisa plates would be washed 3 times by adding 350 µl of wash buffer to the wells and dried on adsorbent paper towels between washes.
5. Biotinylated Human caspase 3 liquid would be now added to each wel
6. The wells would be washed 3 times as described above at step 4.
7. Enzyme conjugate liquid would now be added to the individual wells in the microplate
8. The wells would be washed 3 times as described above at steps 4 and 6 above.
9. Colour reagent (substrate solution) would be added followed by stop solution
10. Optical density would be measured at 450nm using a microplate ELISA reader
11. Values of unknown samples would be read off from the standard curve generated by plotting the optical densities of known standards against their known concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with aneurysmal SAH who are scheduled for surgical or endovascular intervention.
2. Age between 18 to 65 yrs.
3. WFNS grade 1 or 2
4. Fischer grade 1 or 2
5. ASA grade 1 or 2.

Exclusion Criteria:

1. Patients with giant aneurysms of the internal carotid artery that require external carotid-internal carotid bypass or intra operative ligation of internal carotid artery.
2. Patients with known psychiatric disease.
3. Patients with any other neurological or neuro degenerative disorders.
4. History of drug abuse.
5. Patients with any history of carcinoma or any immune deficiency diseases.
6. Intra-operative surgical complications like massive blood loss, prolonged clipping time (>20 minutes), severe intra-operative brain swelling requiring extended craniotomy or lobectomy or precluding replacement of bone flap.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population includes the patients with aneurysmal subarchnoid haemorraghe coming to PGIMER for either supra orbital keyhole approach for aneurysmal clipping or endovascular coiling of the aneurysm
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Estimation of changes in caspase 3 levels as a marker of neurotoxicity in patients with aneurysmal SAH following exposure to general anaesthetics. | baseline( pre- induction), one hour after the exposure to anesthetic agents and after extubation
  enzyme Caspase-3 is used as a marker of apoptosis and will be used as an indirect marker for neurotoxicity caused by general anesthetic agents

CONTACTS AND LOCATIONS:
Overall Officials: MUKILAN BALASUBRAMANIAN, MD, Principal Investigator — PGIMER, chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
since the study is on recruitment phase, it will be decided once the study gets completed